CLINICAL TRIAL: NCT02645318
Title: A Prospective Study of Circulating Tumor DNA Detection by Targeted Sequencing in Surgical Non-Small Cell Lung Cancer Patients
Brief Title: Comparison of Circulating Tumor DNA and Tumor Tissue DNA by Targeted Sequencing in Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: PTHO1501
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Circulating Tumor DNA; Lung cancer; Targeted sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue, peripheral blood cells, and plasma samples were collected from each patient.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Conduct a prospective study to compare gene detection by ctDNA with tumor tissue DNA via targeted DNA sequencing in surgical NSCLC patients.

DETAILED DESCRIPTION:
Previous studies have shown the feasibility of detecting mutation status by circulating tumor DNA (ctDNA)in non-small cell lung cancer (NSCLC) patients. However, no clinical standard method has been established, and most previous studies were lack of prospective clinical data and aimed at advanced NSCLC.

We plan to perform a prospective study including consecutive cases of NSCLC patients who underwent surgical treatments. Primary tumor and plasma samples were collected in each patients and gene mutation analysis were performed immediately after surgery. We utilized the targeted DNA sequencing with a next-generation sequencing (NGS) platform to detect driver somatic mutations in matched tumor DNA (tDNA) and plasma ctDNA samples with matched white blood cell (WBC) DNA as a control. A panel of genes were identified.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is confirmed primary lung cancer by frozen pathologic histology
* Both the fresh tissue tumor and plasma samples are collected for analysis

Exclusion Criteria:

* Patients who received any treatment prior to resection
* Patients who have a history of malignancy
* Paraffin embedded section confirmed small cell lung cancer or unclassified carcinoma
* Tumor specimens where insufficient DNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive cases who were suspected of non-small cell lung cancer and underwent curative-intent resection.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Whether ctDNA can detect genomic alterations in peripheral blood that are consistent with those in matched tumor sample | 2-3 months

SECONDARY OUTCOMES:
Concordance of tDNA and plasma ctDNA gene detection in early stage non-small cell lung cancer | 2-3months
Correlation of ctDNA concentration with clinical features | 2-3months
Comparison of positive predictive value between ctDNA and tumor markers | 2-3months
The relationship between ctDNA concentration and disease free survival(DFS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Chen, M.D., Principal Investigator — Peking University People's Hospital; Jun Wang, M.D., Study Chair — Peking University People's Hospital; Feng Lou, Study Director — San Valley Biotechnology Incorporated
Locations (1):
- Peking University People's Hospital, Beijing, China